CLINICAL TRIAL: NCT04410341
Title: The DPP-4 Inhibitor Vildagliptin as Adjunct in Major Depressive Disorder Patients: A Proof-of-Concept, Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: The DPP-4 Inhibitor Vildagliptin as Adjunct in Major Depressive Disorder Patients
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Institutional and funding constrains
Sponsor: Sadat City University (Other)
Responsible Party: Principal Investigator, Mahmoud Samy Abdallah, Lecturer of Clinical Pharmacy, PhD., Sadat City University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0055/2020
Record Dates: First submitted 2020-05-27; First posted 2020-06-01 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Vildagliptin; Escitalopram

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (Placebo Comparator): Escitalopram 20 mg tablet once daily for 12 week plus placebo tablet once daily for 12 weeks
  Interventions: Drug: Escitalopram 20 mg
- Vildagliptin group (Experimental): Escitalopram 20 mg tablet once daily for 12 week plus Vildagliptin 50mg tablet once daily for 12 weeks
  Interventions: Drug: Vildagliptin 50 MG; Drug: Escitalopram 20 mg

INTERVENTIONS:
Drug: Vildagliptin 50 MG — Vildagliptin, an antidiabetic drug that inhibits the dipeptidyl peptidase- 4 (DPP-4), increases glucagon-like peptide-1 (GLP-1) and regulates blood glucose levels, favoring weight loss and lowering cardiovascular risk.
  Arms: Vildagliptin group
Drug: Escitalopram 20 mg — Escitalopram,Selective serotonin reuptake inhibitor- Cilostazol, a selective phosphodiesterase 3 (PDE3) inhibitor, acts as an antiplatelet agent and has been widely approved for treatment of intermittent claudication with peripheral arterial disease and for secondary prevention of ischemic stroke.

SUMMARY:
Vildagliptin, an antidiabetic drug that inhibits the dipeptidyl peptidase- 4 (DPP-4), increases glucagon-like peptide-1 (GLP-1) and regulates blood glucose levels, favoring weight loss and lowering cardiovascular risk. A retrospective longitudinal study by Rizzo et al. showed that DPP-4 inhibitors administration could have protective effects against cognitive decline in diabetic elderly. Is has been observed that GLP-1 affects brain metabolism, increases neuritic growth, and protects neuronal cells from oxidative stress and death.

ELIGIBILITY:
Inclusion Criteria:

* Eighty adult outpatients with the Diagnostic and Statistical Manual of Mental Disorders-IV (DSM-IV) diagnosis of MDD based on a MINI Neuropsychiatric Interview (MINI) (American Psychiatric Association., 2000; Sheehan et al., 1998), without psychotic features and a total 17 item HAM-D score of at least 18 with item 1 (depressed mood) scored 2 or greater were eligible (Hamilton, 1960).
* Patients were requested to be free of all the psychotropic and anti-inflammatory medications for at least 4 weeks before participating in the study.

Exclusion Criteria:

* Patients with bipolar I or bipolar II disorder
* Patients with personality disorders
* Patients with eating disorders
* Patients with substance dependence or abuse
* Patients with concurrent active medical condition
* Patients with history of seizures
* Patients with history of receiving Electroconvulsive therapy (ECT)
* Patients with inflammatory disorders
* Patients with allergy or contraindications to the used medications
* Patients with finally pregnant or lactating females
* Cardiovascular disorders
* Severe renal impairment: creatinine clearance of ≤ 25 ml/min
* Moderate or severe hepatic impairment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Effect on Hamilton Depression rating scale score (HAM-D score) | 12 week
  The principal measure of the outcome was the 17-items HAM-D. Scoring is based on the 17-item scale and scores of 0-7 are considered as being normal, 8-13 suggest mild depression, 14-17 moderate depression and scores over 17 are indicative of severe depression. Remission is defined as HAM-D total score ≤ 7 (primary outcome). Treatment response is defined as ≥ 50% drop in the HAM-D total score.

SECONDARY OUTCOMES:
Effect on biological markers | Baseline and 12 week
  Serum level of tumor necrosis factor alpha (TNF-α)
Interleukin-6 | Baseline and 12 week
  Serum level of Interleukin-6 (IL-6)
BDNF | Baseline and 12 week
  Serum level of Brain derived neurotrophic factor (BDNF)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Shibīn al Kawm, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF